CLINICAL TRIAL: NCT06723574
Title: Assessing Environmental Sustainability in Urologic Practices: A Systematic Review
Brief Title: Sustainability in Urologic Practices
Acronym: Sustainability
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Collaborators: European Association of Urology Research Foundation (Other)
Responsible Party: Principal Investigator, Selim Soyturk, Principial investigator, Necmettin Erbakan University
Other Study IDs: ResCORE-20
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-12

CONDITIONS: Sustainability in Urologic Practices
Keywords: Sustainability; Urologic Practices; cystoscopy; RIRS; BPH; HoLep; Endourology; reusable; single use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EAU section: EAU section chairs,board members and working group members

SUMMARY:
This research is a two-phase observational study assessing awareness, current practices, barriers, and policy suggestions related to sustainability in urology. The study involves collecting survey data from a broad participant group and conducting a Delphi consensus with experts to develop actionable recommendations.

DETAILED DESCRIPTION:
This study aims to evaluate and promote sustainable practices in urological care by focusing on the environmental impact of urological devices and processes. The study will be conducted in two phases, aiming to assess current practices, challenges, and strategies for reducing the carbon footprint and waste associated with urological procedures, while achieving expert consensus. Participants will include European Association of Urology (EAU) section chairs and board members, ensuring comprehensive analyses and authoritative recommendations.

In the first phase, an online survey will be administered to 150-200 participants. The survey will be distributed via platforms such as Google Forms or Qualtrics and will collect data on awareness, current practices, and challenges related to the environmental sustainability of urological devices. These findings will serve as the foundation for the Delphi consensus process in the second phase.

In the second phase, a Delphi panel consisting of 12-15 experts nominated from EAU sections will conduct a structured consensus process. This process will include three rounds:

1. Round 1: Open-ended questions will be used to gather expert opinions based on the findings of the survey.
2. Round 2: Proposed strategies will be evaluated and prioritized by the panel.
3. Round 3: Consensus will be reached on actionable recommendations for sustainable practices.

Participation in the study will be entirely voluntary, and informed consent will be obtained from all participants. All data collected during the survey and Delphi processes will be anonymized and used solely for the purposes of the study. Data will be handled in compliance with the General Data Protection Regulation (GDPR) and applicable local data protection laws.

ELIGIBILITY:
Inclusion Criteria:

* EAU Section Chairs and Board Members
* Individuals who voluntarily agree to participate in the study.

Exclusion Criteria:

* Individuals who refuse to participate in the study.
* Individuals who do not provide the required information or complete the survey incompletely.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 200 Participants
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Consensus on Sustainable Practices in Urology | Within 6 months of initiating the Delphi process.
  The number of sustainable practices identified and agreed upon by the Delphi panel (consensus defined as ≥70% agreement among panelists). Measure Type: Binary (Consensus Achieved/Not Achieved).
Awareness and Current Practices Score | At the completion of the online survey phase (approximately 3 months after the study begins).
  Mean score from the online survey evaluating participants' awareness of environmental sustainability in urology and current sustainable practices (measured on a 5-point Likert scale). Measure Type: Continuous (score range: 1-5).

SECONDARY OUTCOMES:
Identified Barriers to Sustainable Practices | Within 3 months of survey completion.
  The percentage of participants identifying specific barriers to implementing sustainable practices in their institutions (categorized into themes such as cost, lack of awareness, or technical challenges).Categorical (number of barriers per theme).

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

REFERENCES:
- [Background] Elliott CS. Sustainability in Urology: Single-use Versus Reusable Catheters for Intermittent Catheterization. Eur Urol Focus. 2023 Nov;9(6):888-890. doi: 10.1016/j.euf.2023.09.012. Epub 2023 Oct 4. PMID 37802716
- [Background] Baboudjian M, Pradere B, Martin N, Gondran-Tellier B, Angerri O, Boucheron T, Bastide C, Emiliani E, Misrai V, Breda A, Lechevallier E. Life Cycle Assessment of Reusable and Disposable Cystoscopes: A Path to Greener Urological Procedures. Eur Urol Focus. 2023 Jul;9(4):681-687. doi: 10.1016/j.euf.2022.12.006. Epub 2022 Dec 20. PMID 36543725
- [Background] Misrai V, Rijo E, Cottenceau JB, Zorn KC, Enikeev D, Elterman D, Bhojani N, De La Taille A, Herrmann TRW, Robert G, Pradere B. A Standardized Method for Estimating the Carbon Footprint of Disposable Minimally Invasive Surgical Devices: Application in Transurethral Prostate Surgery. Ann Surg Open. 2021 Sep 7;2(3):e094. doi: 10.1097/AS9.0000000000000094. eCollection 2021 Sep. PMID 37635829
- [Derived] Tozsin A, Ahmed K, Soyturk S, Pradere B, Dasgupta P, Sonmez MG, Keller EX, Omar MI, Mallet R, Aydin A, Gadzhiev N, Cakir OO, Vasquez JL, Akgul B, Arslan E, Silay SM, Sanguedolce F, Roupret M, Musquera M, Ralph D, Colecchia M, Finazzi Agro E, Bettocchi C, Traxer O, Tunc L, Rassweiler J, Herrmann TRW, Knoll T, Guven S. Achieving sustainability in urology: a consensus study by the European association of urology (EAU) section office. World J Urol. 2025 Nov 15;43(1):697. doi: 10.1007/s00345-025-06084-4. PMID 41240108